CLINICAL TRIAL: NCT01312909
Title: A Twelve-week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study With Follow-up Evaluating The Safety And Efficacy Of Varenicline For Smoking Cessation In Healthy Adolescent Smokers
Brief Title: Smoking Cessation Study In Healthy Adolescent Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3051073; CHANTIX (Other: Alias Study Number)
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Smoking Cessation
Keywords: smoking cessation in adolescents
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Varenicline 1mg BID (Experimental): Oral Varenicline 1mg BID, or 1/2 that dose (0.5mg BID) for those subjects that weigh less than or equal to 55kg at baseline, for twelve weeks, follow-up through Week 52
  Interventions: Drug: Varenicline 1mg BID
- Varenicline 0.5mg BID (Experimental): Oral Varenicline 0.5mg BID, or 1/2 that dose (0.5 QD) for those subjects that weigh less than or equal to 55kg at baseline, for twelve weeks, follow-up through Week 52
  Interventions: Drug: Varenicline 0.5mg BID
- Placebo (Placebo Comparator): Oral placebo for twelve weeks,follow-up through Week 52
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline 1mg BID — Oral Varenicline 1mg BID, or 1/2 that dose (0.5mg BID) for those subjects that weigh less than or equal to 55kg at baseline, for twelve weeks, follow-up through Week 52
  Arms: Varenicline 1mg BID
Drug: Varenicline 0.5mg BID — Oral Varenicline 0.5mg BID, or 1/2 that dose (0.5 QD) for those subjects that weigh less than or equal to 55kg at baseline, for twelve weeks, follow-up through Week 52
  Arms: Varenicline 0.5mg BID
Drug: Placebo — Oral placebo for twelve weeks,follow-up through Week 52
  Arms: Placebo

SUMMARY:
The study is designed to see if varenicline combined with age appropriate (adolescent) smoking cessation counseling will help teens quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 12 and 19, inclusive.
* Subjects smoking at least an average of 5 cigarettes per day, motivated to stop smoking,
* Subjects must have at least one prior failed attempt to quit smoking.

Exclusion Criteria:

* Subjects with history, current diagnosis, or treatment of major depression disorder, anxiety disorders, panic disorder, hostility or aggression disorder, perceptual/thinking disturbances, mania, psychosis, bipolar disorder, personality disorder, eating disorder or severe emotional problems (in the past year).
* Subjects with a prior suicide attempt: subjects hospitalized within the past 12 months due to suicidal ideation or suicidal behavior; subjects considered to have serious suicidal ideation or suicidal behavior in the past 12 months; active suicidal ideation or behavior identified at the screening or baseline visit.
* Evidence of alcohol and substance abuse/dependence (other than nicotine) within 3 months prior to screening.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 312 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (79):
- United States (56):
  - IICR, Inc. (DBA: International Institute of Clinical Research), Ozark, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Omega Clinical Trials, LLC, La Habra, California
  - Synergy Clinical Research Center, National City, California
  - Pacific Research Partners, LLC, Oakland, California
  - North County Clinical Research, Oceanside, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Western Affiliated Research Institute, Denver, Colorado
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale University, SATU, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Avail Clinical Research, LLC, DeLand, Florida
  - Hope Clinical Research, Kissimmee, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - L & L Research Choices, Miami, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Comprehensive Clinical Development Inc., St. Petersburg, Florida
  - Barney Greenspan, Ph.D, Meridian, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Midwest Behavioral Health, Evansville, Indiana
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Pedia Research, LLC, Newburgh, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Louisiana Research Associates, Inc, New Orleans, Louisiana
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Psychiatric Care & Research Center, O'Fallon, Missouri
  - Mid-America Clinical Research, LLC, St Louis, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Wake Internal Medicine Consultants, Inc, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Insite Clinical Research, LLC, DeSoto, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Thomas Murray DeMoor, MD, San Antonio, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Zain Research, LLC, Richland, Washington
  - Dean Foundation for Health Research and Education, Middleton, Wisconsin
- Canada (3):
  - Kids Clinic, Ajax, Ontario
  - Private Practice of Robert J. Camargo, Newmarket, Ontario
  - SKDS Research Inc., Newmarket, Ontario
- LTD" Rustavi Psychological Health Center", Rustavi, Georgia
- Russia (9):
  - Leningrad Regional Dispensary of Narcology, Village Novoe Devyatkino, Leningradskaya Oblast'
  - GBUZ City childrens out-patient clinic # 10 of Moscow, Moscow
  - GOBUZ Murmansk Regional Narcology Dispensary, Murmansk
  - LLC City Neurological Center "Sibneuromed", Novosibirsk
  - LLC " Alliance Biomedical - Russian Group", Saint Petersburg
  - LLC Medical Technologies, Saint Petersburg
  - FSBI V.M.Bekhterev National Research Medical Center for Psychiatry and Neurology of RF MoH, Saint Petersburg
  - First St. Petersburg State Medical University, Saint Petersburg
  - GBUZ Samara Regional Childrens Health camp Yunost, Samara
- South Korea (4):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea St. Vincent Hospital, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Hospital, Daegu
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Fediuk DJ, Sweeney K, Sahasrabudhe V, McRae T, Byon W. Population pharmacokinetics and exposure-response analyses of varenicline in adolescent smokers. CPT Pharmacometrics Syst Pharmacol. 2021 Jul;10(7):769-781. doi: 10.1002/psp4.12645. Epub 2021 Jun 17. PMID 34062053
- [Derived] Gray KM, Rubinstein ML, Prochaska JJ, DuBrava SJ, Holstein AR, Samuels L, McRae TD. High-dose and low-dose varenicline for smoking cessation in adolescents: a randomised, placebo-controlled trial. Lancet Child Adolesc Health. 2020 Nov;4(11):837-845. doi: 10.1016/S2352-4642(20)30243-1. Epub 2020 Sep 25. PMID 32979939
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051073&StudyName=Smoking%20Cessation%20Study%20In%20Healthy%20Adolescent%20Smokers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 3 phases: Screening (3 weeks before first dose of study drug); treatment (from Week 2 to Week 12 after a 2-week titration) and non-treatment follow-up (Week 13 through Week 52).
Groups:
- Varenicline High Dose: Participants received 2 tablets of Varenicline 0.5 milligram (mg) (total dose 1 mg) orally, twice daily from Week 2 to Week 12 after a 2-week titration. Participants with a body weight less than or equal to (<=) 55 kilograms (kg) had Varenicline dose reduced by half, and received one tablet of Varenicline 0.5 mg and one matching placebo tablet orally, twice daily from Week 2 to Week 12 after a 2-week titration.
- Varenicline Low Dose: Participants received one tablet of Varenicline 0.5 mg and one matching placebo tablet orally, twice daily from Week 2 to Week 12 after a 2-week titration. Participants with a body weight <= 55 kg had Varenicline dose reduced by half and received one tablet of Varenicline 0.5 mg and one matching placebo tablet orally, in the morning and 2 tablets of matching placebo orally, in the evening from Week 2 to Week 12 after a 2-week titration.
- Placebo: Participants received 2 tablets of placebo (matched to Varenicline) orally, twice daily from Week 2 to Week 12 after a 2-week titration.
Period: Overall Study
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Started | 109 | 103 | 100
Treated | 108 | 100 | 99
Completed | 67 | 67 | 53
Not Completed | 42 | 36 | 47
Not completed — Randomized but not treated | 1 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 3
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Other | 9 | 6 | 11
Not completed — Withdrawal by Subject | 8 | 10 | 7
Not completed — Lost to Follow-up | 21 | 17 | 20
Not completed — Insufficient clinical response | 0 | 0 | 1
Not completed — Entrance criteria not met | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who took at least one dose of randomized study medication, including partial doses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo | Total
Number analyzed (Participants) | 108 | 100 | 99 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (2.0) | 16.0 (1.7) | 15.8 (1.8) | 15.9 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 36 | 111
  Male | 70 | 63 | 63 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 81 | 73 | 74 | 228
  Black | 9 | 9 | 5 | 23
  Asian | 16 | 18 | 19 | 53
  Other | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: 4-Week Continuous Abstinence Rate: Percentage of Participants Who Remained Abstinent From Week 9 Through Week 12
Description: The percentage of participants who, at each visit from Week 9 through Week 12, reported no smoking and no use of other nicotine-containing products since the last study visit (on the Nicotine Use Inventory) and at each of these visits were confirmed to have quit based on urine cotinine less than 200 nanograms/milliliter (ng/mL).
Time Frame: Week 9 through Week 12
Population: The full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 109 | 103 | 100
percentage of participants | 20.2 | 27.2 | 18.0
Statistical Analysis 1: Comparison: Varenicline High Dose vs Placebo; Odds ratios and p-values were obtained from a logistic regression model with terms treatment, age strata, body weight strata and pooled center. A testing order was used to control type I error. 1mg Varenicline twice daily group was tested against placebo first, and if statistically significant difference was observed, the 0.5 mg Varenicline twice daily group was tested against placebo; Test type: Superiority; p = 0.6337, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.59 to 2.37]
Statistical Analysis 2: Comparison: Varenicline Low Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1114, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.88 to 3.39]

2. Secondary Outcome: Percentage of Participants With 7-Day Point Prevalence of Smoking Abstinence at Weeks 12, 24 and 52
Description: The percentage of participants who reported no smoking and no use of other nicotine-containing products (treatment phase) or tobacco products (non-treatment phase) on the Nicotine Use Inventory in the 7 days prior to the study visits or telephone contacts at Week 12,24 and 52.
Time Frame: Weeks 12, 24 and 52
Population: The full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 109 | 103 | 100
percentage of participants
  Week 12 | 31.2 | 37.9 | 23.0
  Week 24 | 31.2 | 35.9 | 23.0
  Week 52 | 28.4 | 35.0 | 20.0
Statistical Analysis 1: Comparison: Varenicline High Dose vs Placebo; Week 12; Test type: Superiority; p = 0.5793, Regression, Logistic; Odds ratios and p-values were obtained from separate logistic regression models of treatment, pooled center, age strata and body weight strata; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.62 to 2.38]
Statistical Analysis 2: Comparison: Varenicline Low Dose vs Placebo; Week 12; Test type: Superiority; p = 0.0932, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.91 to 3.51]
Statistical Analysis 3: Comparison: Varenicline High Dose vs Placebo; Week 24; Test type: Superiority; p = 0.5647, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.61 to 2.50]
Statistical Analysis 4: Comparison: Varenicline Low Dose vs Placebo; Week 24; Test type: Superiority; p = 0.2917, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.72 to 2.96]
Statistical Analysis 5: Comparison: Varenicline High Dose vs Placebo; Week 52; Test type: Superiority; p = 0.5616, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.58 to 2.69]
Statistical Analysis 6: Comparison: Varenicline Low Dose vs Placebo; Week 52; Test type: Superiority; p = 0.1300, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.84 to 3.78]

3. Secondary Outcome: Daily Number of Cigarettes Smoked at Baseline
Description: The average number of cigarettes smoked per day in the past 7 days reported at the baseline visit.
Time Frame: Baseline
Population: The full analysis set included all randomized participants.
Measure: Mean (Standard Error); unit: cigarettes smoked per day
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 109 | 103 | 100
cigarettes smoked per day | 10.68 (0.624) | 9.56 (0.530) | 9.57 (0.531)

4. Secondary Outcome: Change From Baseline in Daily Number of Cigarettes Smoked at Weeks 12, 24, and 52
Description: The reduction in the number of the cigarettes smoked was calculated by subtracting the reported average number of cigarettes smoked per day in the past 7 days at Weeks 12, 24 and 52 from the average number of cigarettes smoked per day in the past 7 days reported at the baseline visit.
Time Frame: Baseline, Weeks 12, 24, and 52
Population: The full analysis set included all randomized participants. The longitudinal model included all participants regardless of observed visits.
Measure: Least Squares Mean (Standard Error); unit: cigarettes smoked per day
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 109 | 103 | 100
cigarettes smoked per day
  Change at Week 12 | -8.56 (0.43) | -8.20 (0.44) | -8.01 (0.46)
  Change at Week 24 | -6.93 (0.44) | -7.31 (0.45) | -6.59 (0.48)
  Change at Week 52 | -6.80 (0.45) | -7.74 (0.46) | -6.98 (0.48)
Statistical Analysis 1: Comparison: Varenicline High Dose vs Placebo; Week 12: Analysis was performed using longitudinal repeated measures model with the change from baseline average number of Cigarettes Smoked as the dependent variable, including terms treatment, visit, age strata, body weight strata, pooled center, baseline measure and treatment by visit interaction; Test type: Superiority; p = 0.3540, Longitudinal repeated measures model; Least square (LS) mean difference = -0.54, 95% CI 2-sided [-1.69 to 0.60], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: Varenicline Low Dose vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7574, Longitudinal repeated measures model; LS mean difference = -0.18, 95% CI 2-sided [-1.35 to 0.98], Standard Error of Mean 0.59
Statistical Analysis 3: Comparison: Varenicline High Dose vs Placebo; Week 24: Analysis was performed using longitudinal repeated measures model with the change from baseline average number of Cigarettes Smoked as the dependent variable, including terms treatment, visit, age strata, body weight strata, pooled center, baseline measure and treatment by visit interaction; Test type: Superiority; p = 0.5676, Longitudinal repeated measures model; LS mean difference = -0.34, 95% CI 2-sided [-1.53 to 0.84], Standard Error of Mean 0.60
Statistical Analysis 4: Comparison: Varenicline Low Dose vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.2356, Longitudinal repeated measures model; LS mean difference = -0.72, 95% CI 2-sided [-1.92 to 0.47], Standard Error of Mean 0.61
Statistical Analysis 5: Comparison: Varenicline High Dose vs Placebo; Week 52: Analysis was performed using longitudinal repeated measures model with the change from baseline average number of Cigarettes Smoked as the dependent variable, including terms treatment, visit, age strata, body weight strata, pooled center, baseline measure and treatment by visit interaction; Test type: Superiority; p = 0.7730, Longitudinal repeated measures model; LS mean difference = 0.18, 95% CI 2-sided [-1.03 to 1.38], Standard Error of Mean 0.62
Statistical Analysis 6: Comparison: Varenicline Low Dose vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.2166, Longitudinal repeated measures model; LS mean difference = -0.77, 95% CI 2-sided [-1.99 to 0.45], Standard Error of Mean 0.62

5. Secondary Outcome: Continuous Abstinence Rate: Percentage of Participants Who Remained Abstinent From Week 9 Through Week 24 and Week 52
Description: The percentage of participants who, at each visit from Week 9 to 52 (inclusive), reported no smoking and no use of other nicotine-containing products (Weeks 9-12) or tobacco products (Weeks 13-52) since the last study visit/last contact (on the Nicotine Use Inventory) and at any of the study visits were confirmed to have quit based on urine cotinine less than 200 ng/mL.
Time Frame: Week 9 through Week 24; Week 9 through Week 52
Population: The full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 109 | 103 | 100
percentage of participants
  Week 9 through Week 24 | 10.1 | 24.3 | 13.0
  Week 9 through Week 52 | 8.3 | 20.4 | 9.0
Statistical Analysis 1: Comparison: Varenicline High Dose vs Placebo; Week 9 through Week 24: Odds ratios and p-values were obtained from a logistic regression model including the main effects of treatment, pooled center, age strata and body weight strata; Test type: Superiority; p = 0.6133, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.34 to 1.90]
Statistical Analysis 2: Comparison: Varenicline Low Dose vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0335, Regression, Logistic; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.07 to 4.79]
Statistical Analysis 3: Comparison: Varenicline High Dose vs Placebo; Week 9 through Week 52: Odds ratios and p-values were obtained from a logistic regression model including the main effects of treatment, pooled center, age strata and body weight strata; Test type: Superiority; p = 0.9874, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.37 to 2.65]
Statistical Analysis 4: Comparison: Varenicline Low Dose vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0188, Regression, Logistic; Odds Ratio (OR) = 2.79, 95% CI 2-sided [1.19 to 6.55]

6. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both non-serious AEs and SAEs.
Time Frame: First dose up to last dose (up-to Week 12) plus 30 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 108 | 100 | 99
Participants | 65 | 53 | 52

7. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent were events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to drug Varenicline was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category. An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both non-serious AEs and SAEs.
Time Frame: First dose up to last dose (up-to Week 12) plus 30 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 108 | 100 | 99
Participants | 46 | 28 | 27

8. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Neuropsychiatric Adverse Event Elicited by Neuropsychiatric Adverse Event Interview (NAEI)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE: AE causing: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent/significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Solicited AEs collected by semi-structured NAEI inquiring about AEs: depression, anxiety, delusions, hallucinations, paranoia, psychosis, mania, panic, agitation, dissociative states, feeling abnormal, hostility, aggression and homicidal ideation. If a participant had a positive response to any item on the NAEI, investigator determined if it met criteria AE criteria.
Time Frame: First dose up to last dose (up-to Week 12) plus 30 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 108 | 100 | 99
Participants
  Neuropsychiatric AEs | 18 | 11 | 12
  Neuropsychiatric SAEs | 0 | 0 | 0

9. Other Pre Specified Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories);was an interview-based instrument to systematically assess suicidal ideation and suicidal behavior.C-SSRS assessed whether participant experienced any of the following:completed suicide;suicide attempt(response of "Yes" on "actual attempt");preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior","aborted attempt" or "interrupted attempt"),suicidal ideation ("Yes" on "wish to be dead","non-specific active suicidal thoughts","active suicidal ideation with methods without intent to act or some intent to act,without specific plan or with specific plan and intent,any self-injurious behavior with no suicidal intent ("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").Here,number of participants with positive response (response of "yes") to suicidal behavior or/and Ideation,any non-suicidal self-injurious behavior were reported.
Time Frame: Screening, Baseline, Week 1 up to Week 12 (treatment-emergent [TE]), thereafter up to Week 52 (last follow-up [FU])
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 108 | 100 | 99
Participants
  Screening:Suicidal Behavior or/and Ideation | 2 | 3 | 2
  Screening:Suicidal Ideation | 2 | 3 | 2
  Screening: Wish to be Dead | 2 | 2 | 2
  Screening: Non-Specific Active Suicidal Thoughts | 1 | 1 | 2
  Screen:Self Injurious Behavior, no Suicidal Intent | 3 | 3 | 2
  TE:Suicidal Behavior or/and Ideation: number analyzed (Participants) | 105 | 99 | 96
  TE:Suicidal Behavior or/and Ideation | 1 | 0 | 1
  TE:Suicidal Ideation: number analyzed (Participants) | 105 | 99 | 96
  TE:Suicidal Ideation | 1 | 0 | 1
  TE: Wish to be Dead: number analyzed (Participants) | 105 | 99 | 96
  TE: Wish to be Dead | 1 | 0 | 1
  TE: Non-Specific Active Suicidal Thoughts: number analyzed (Participants) | 105 | 99 | 96
  TE: Non-Specific Active Suicidal Thoughts | 0 | 0 | 1
  TE:Self Injurious Behavior, no Suicidal Intent | 0 | 0 | 1

10. Other Pre Specified Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) - Anxiety (HADS-A) Total Scores at Specified Time-points
Description: The HADS is a self-administered questionnaire measuring anxiety. Hospital Anxiety and Depression Scale Anxiety subscale (HADS-A) consisted of 7 items that were assessed on a scale of 0 = no anxiety to 3 = severe feeling of anxiety. Total HADS-A subscale score range from 0 = no anxiety to 21 = severe anxiety; higher scores indicated more severe anxiety.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 20, 28, 36, 44, and 52
Population: The safety analysis set included all participants who took at least one dose of randomized study medication, including partial doses. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 108 | 100 | 99
units on a scale
  Baseline | 2.4 (2.05) | 1.9 (2.06) | 2.3 (2.26)
  Change at Week 1: number analyzed (Participants) | 104 | 99 | 94
  Change at Week 1 | -0.6 (1.86) | -0.5 (1.53) | -0.3 (1.91)
  Change at Week 2: number analyzed (Participants) | 102 | 97 | 89
  Change at Week 2 | -1.1 (1.95) | -0.7 (1.90) | -0.5 (2.18)
  Change at Week 3: number analyzed (Participants) | 101 | 91 | 87
  Change at Week 3 | -1.2 (1.85) | -0.8 (1.96) | -1.0 (2.09)
  Change at Week 4: number analyzed (Participants) | 95 | 88 | 87
  Change at Week 4 | -1.5 (1.83) | -0.9 (2.31) | -0.9 (2.21)
  Change at Week 5: number analyzed (Participants) | 92 | 86 | 81
  Change at Week 5 | -1.3 (2.03) | -1.0 (2.12) | -1.2 (2.19)
  Change at Week 6: number analyzed (Participants) | 90 | 84 | 75
  Change at Week 6 | -1.5 (1.91) | -1.0 (2.25) | -1.2 (2.31)
  Change at Week 7: number analyzed (Participants) | 88 | 79 | 73
  Change at Week 7 | -1.6 (2.13) | -1.1 (2.41) | -1.2 (2.39)
  Change at Week 8: number analyzed (Participants) | 88 | 81 | 74
  Change at Week 8 | -1.5 (2.11) | -1.1 (2.20) | -1.3 (1.99)
  Change at Week 9: number analyzed (Participants) | 86 | 77 | 69
  Change at Week 9 | -1.4 (2.17) | -1.2 (2.35) | -1.1 (2.13)
  Change at Week 10: number analyzed (Participants) | 81 | 80 | 70
  Change at Week 10 | -1.4 (2.07) | -1.2 (2.44) | -1.1 (2.34)
  Change at Week 11: number analyzed (Participants) | 83 | 80 | 67
  Change at Week 11 | -1.4 (2.00) | -1.2 (2.23) | -1.3 (2.12)
  Change at Week 12: number analyzed (Participants) | 82 | 77 | 65
  Change at Week 12 | -1.4 (2.07) | -1.3 (2.31) | -1.2 (2.15)
  Change at Week 13: number analyzed (Participants) | 84 | 76 | 65
  Change at Week 13 | -1.5 (2.13) | -1.2 (2.17) | -1.2 (2.33)
  Change at Week 14: number analyzed (Participants) | 79 | 76 | 62
  Change at Week 14 | -1.4 (2.33) | -1.2 (2.53) | -1.2 (2.19)
  Change at Week 15: number analyzed (Participants) | 76 | 74 | 62
  Change at Week 15 | -1.7 (2.09) | -1.3 (2.43) | -1.0 (3.35)
  Change at Week 16: number analyzed (Participants) | 76 | 74 | 61
  Change at Week 16 | -1.6 (2.16) | -1.2 (2.44) | -1.1 (2.54)
  Change at Week 20: number analyzed (Participants) | 78 | 72 | 60
  Change at Week 20 | -1.5 (2.28) | -1.2 (2.31) | -1.3 (2.21)
  Change at Week 28: number analyzed (Participants) | 72 | 69 | 56
  Change at Week 28 | -1.5 (2.54) | -1.2 (2.46) | -1.2 (2.38)
  Change at Week 36: number analyzed (Participants) | 72 | 67 | 53
  Change at Week 36 | -1.4 (2.42) | -1.2 (2.51) | -1.3 (2.03)
  Change at Week 44: number analyzed (Participants) | 70 | 66 | 53
  Change at Week 44 | -1.8 (2.21) | -1.2 (2.34) | -1.0 (1.90)
  Change at Week 52: number analyzed (Participants) | 67 | 67 | 53
  Change at Week 52 | -1.6 (2.20) | -1.1 (2.39) | -1.5 (2.06)

11. Other Pre Specified Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Scores - Depression Total Score at Specified Time-Points
Description: Hospital Anxiety and Depression Scale Depression subscale (HADS-D) consists of 7 items that were assessed on a scale of 0 = no depression to 3 = severe feeling of depression. Total HADS-D subscale score range from 0 = no depression to 21 = severe feeling of depression; higher scores indicated a greater intensity of depression.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 20, 28, 36, 44, and 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 108 | 100 | 99
units on a scale
  Baseline | 1.5 (1.93) | 1.4 (1.79) | 1.4 (1.83)
  Change at Week 1: number analyzed (Participants) | 104 | 99 | 94
  Change at Week 1 | -0.4 (1.43) | -0.2 (1.18) | 0.1 (1.61)
  Change at Week 2: number analyzed (Participants) | 102 | 97 | 89
  Change at Week 2 | -0.5 (1.57) | -0.2 (1.65) | -0.1 (1.80)
  Change at Week 3: number analyzed (Participants) | 101 | 91 | 87
  Change at Week 3 | -0.5 (1.39) | -0.3 (1.55) | -0.3 (1.79)
  Change at Week 4: number analyzed (Participants) | 95 | 88 | 87
  Change at Week 4 | -0.7 (1.39) | -0.3 (1.79) | -0.4 (2.00)
  Change at Week 5: number analyzed (Participants) | 92 | 86 | 81
  Change at Week 5 | -0.6 (1.66) | -0.3 (1.97) | -0.3 (1.88)
  Change at Week 6: number analyzed (Participants) | 90 | 84 | 75
  Change at Week 6 | -0.6 (1.85) | -0.4 (1.60) | -0.5 (1.83)
  Change at Week 7: number analyzed (Participants) | 88 | 79 | 73
  Change at Week 7 | -0.7 (1.52) | -0.5 (1.91) | -0.4 (2.13)
  Change at Week 8: number analyzed (Participants) | 88 | 81 | 74
  Change at Week 8 | -0.8 (1.87) | -0.5 (1.80) | -0.5 (1.80)
  Change at Week 9: number analyzed (Participants) | 86 | 77 | 69
  Change at Week 9 | -0.8 (1.63) | -0.5 (1.85) | -0.5 (2.30)
  Change at Week 10: number analyzed (Participants) | 81 | 80 | 70
  Change at Week 10 | -0.9 (1.67) | -0.7 (1.63) | -0.4 (2.77)
  Change at Week 11: number analyzed (Participants) | 83 | 80 | 67
  Change at Week 11 | -0.7 (1.53) | -0.9 (1.66) | -0.5 (2.11)
  Change at Week 12: number analyzed (Participants) | 82 | 77 | 65
  Change at Week 12 | -0.7 (1.79) | -0.7 (1.72) | -0.6 (2.11)
  Change at Week 13: number analyzed (Participants) | 84 | 76 | 65
  Change at Week 13 | -0.6 (2.16) | -0.7 (1.79) | -0.7 (1.95)
  Change at Week 14: number analyzed (Participants) | 79 | 76 | 62
  Change at Week 14 | -0.8 (1.96) | -0.6 (1.84) | -0.5 (2.22)
  Change at Week 15: number analyzed (Participants) | 76 | 74 | 62
  Change at Week 15 | -0.8 (1.83) | -0.8 (1.84) | -0.3 (3.26)
  Change at Week 16: number analyzed (Participants) | 76 | 74 | 61
  Change at Week 16 | -0.6 (2.09) | -0.6 (2.08) | -0.2 (2.79)
  Change at Week 20: number analyzed (Participants) | 78 | 72 | 60
  Change at Week 20 | -0.8 (1.71) | -0.8 (1.84) | -0.6 (2.24)
  Change at Week 28: number analyzed (Participants) | 72 | 69 | 56
  Change at Week 28 | -0.9 (1.63) | -0.8 (1.90) | -0.5 (2.40)
  Change at Week 36: number analyzed (Participants) | 72 | 67 | 53
  Change at Week 36 | -0.7 (2.19) | -0.8 (1.77) | -0.4 (2.40)
  Change at Week 44: number analyzed (Participants) | 70 | 66 | 53
  Change at Week 44 | -0.9 (1.93) | -0.9 (1.78) | -0.3 (2.44)
  Change at Week 52: number analyzed (Participants) | 67 | 67 | 53
  Change at Week 52 | -0.7 (1.81) | -0.8 (1.67) | -0.6 (2.02)

12. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory abnormalities: Lymphocytes Absolute (Abs), Lymphocytes percentage (%), Total Neutrophils (Abs), Neutrophils %: <0.8*LLN or >1.2*ULN; Basophils (Abs), Basophils %Eosinophils (Abs), Eosinophils %, Monocytes (Abs), Monocytes %:> 1.2*ULN; Total Bilirubin milligram per deciliter (mg/dl) >1.5*ULN; alanine aminotransferase: >3.0*ULN; Blood urea nitrogen, Creatinine: >1.3*ULN; Uric acid :> 1.2*ULN.
Time Frame: Baseline up to Week 12
Population: The safety analysis set included all participants who took at least one dose of randomized study medication, including partial doses. Here, 'Number of Participants Analyzed= participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 103 | 93 | 90
Participants | 35 | 33 | 26

13. Other Pre Specified Outcome: Change From Baseline in Blood Pressure (BP) at Week 12
Description: Measurement of BP included supine and sitting systolic BP, standing systolic BP, supine and sitting diastolic BP and standing diastolic BP. Blood pressure was taken after participants rested in a sitting position for 5 minutes. BP was recorded after participants had been supine for approximately 5 minutes, and then orthostatic blood pressure was recorded immediately when the participant stood.
Time Frame: Baseline, Week 12
Population: The safety analysis set included all participants who took at least one dose of randomized study medication, including partial doses. Here, 'Number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: millimeters of mercury (mmHg)
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 77 | 77 | 59
millimeters of mercury (mmHg)
  Supine Systolic BP:Baseline | 115.0 [85 to 164] | 114.0 [92 to 136] | 109.0 [95 to 142]
  Supine Systolic BP:Change at Week 12 | 0.0 [-33 to 25] | 0.0 [-32 to 31] | 0.0 [-35 to 43]
  Sitting Systolic BP:Baseline | 117.0 [90 to 148] | 115.0 [95 to 139] | 113.0 [95 to 135]
  Sitting Systolic BP:Change at Week 12 | -1.0 [-24 to 31] | 0.0 [-30 to 28] | 2.0 [-28 to 28]
  Standing Systolic BP:Baseline | 116.0 [88 to 157] | 115.0 [92 to 155] | 112.0 [90 to 136]
  Standing Systolic BP:Change at Week 12 | 0.0 [-30 to 40] | 0.0 [-21 to 53] | 3.0 [-18 to 47]
  Supine Diastolic BP:Baseline | 69.0 [45 to 99] | 66.0 [45 to 84] | 65.0 [50 to 90]
  Supine Diastolic BP:Change at Week 12 | 0.0 [-26 to 17] | 0.0 [-20 to 22] | 0.0 [-35 to 21.0]
  Sitting Diastolic BP:Baseline | 72.0 [50 to 94] | 70.0 [38 to 92] | 69.0 [47 to 87]
  Sitting Diastolic BP:Change at Week 12 | 0.0 [-20 to 28] | -1.0 [-35 to 23] | 1.0 [-18 to 22]
  Standing Diastolic BP:Baseline | 73.0 [57 to 106] | 72.0 [55 to 99] | 70.0 [50 to 92]
  Standing Diastolic BP:Change at Week 12 | 0.0 [-28 to 22] | -1.0 [-43 to 23] | 2.0 [-21 to 20]

14. Other Pre Specified Outcome: Change From Baseline in Pulse Rate at Week 12
Description: Measurement of pulse rate included supine, sitting and standing pulse rate. Pulse rate was taken after participants rested in a sitting position for 5 minutes. Pulse rate was recorded after participants had been supine for approximately 5 minutes and then immediately upon standing.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Median (Full Range); unit: beats per minute (bpm)
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
Number analyzed (Participants) | 77 | 77 | 59
beats per minute (bpm)
  Supine Pulse Rate:Baseline | 75.0 [50 to 111] | 72.0 [50 to 105] | 72.0 [54 to 113]
  Supine Pulse Rate:Change at Week 12 | 0.0 [-32 to 44] | 1.0 [-23 to 23] | 3.0 [-30 to 29]
  Sitting Pulse Rate:Baseline | 75.0 [58 to 118] | 75.0 [48 to 113] | 77.0 [58 to 115]
  Sitting Pulse Rate:Change at Week 12 | -1.0 [-22 to 25] | 0.0 [-33 to 30] | 1.0 [-43 to 36]
  Standing Pulse Rate:Baseline | 84.0 [61 to 139] | 85.0 [61 to 119] | 85.0 [63 to 122]
  Standing Pulse Rate:Change at Week 12 | 1.0 [-35 to 44] | -3.0 [-25 to 32] | -3.0 [-53 to 44]

ADVERSE EVENTS:
Time Frame: First dose up to last dose (up-to Week 12) plus 30 days
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Varenicline High Dose | Varenicline Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 3/108 | 1/100 | 1/99
Other Adverse Events (participants affected / at risk) | 65/108 | 53/100 | 51/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline High Dose (N=108) | Varenicline Low Dose (N=100) | Placebo (N=99)
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 1
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline High Dose (N=108) | Varenicline Low Dose (N=100) | Placebo (N=99)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 26 | 19 | 12
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 14 | 2 | 2
Asthenia (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Feeling jittery (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 2 | 1
Multiple allergies (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Gonorrhoea (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3 | 5
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 3 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 3 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 3 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0
Blood pressure orthostatic decreased (Investigations) | 0 | 1 | 1
Body mass index increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 7 | 3
Dysgeusia (Nervous system disorders) | 1 | 3 | 2
Headache (Nervous system disorders) | 14 | 5 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 2 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Sleep paralysis (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 2
Tremor (Nervous system disorders) | 1 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 8 | 5 | 4
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 9 | 5 | 5
Anxiety (Psychiatric disorders) | 6 | 4 | 7
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1
Aversion (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 2 | 0
Depression (Psychiatric disorders) | 3 | 2 | 3
Dissociation (Psychiatric disorders) | 0 | 1 | 0
Flat affect (Psychiatric disorders) | 1 | 0 | 1
Grief reaction (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 2
Hostility (Psychiatric disorders) | 7 | 3 | 4
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Irritability (Psychiatric disorders) | 2 | 3 | 1
Mania (Psychiatric disorders) | 1 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2012-07-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT01312909/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT01312909/SAP_001.pdf